CLINICAL TRIAL: NCT05776264
Title: Exercise Strategies to Motivate and Relieve Stress in Adults With Chronic Cardiopulmonary Conditions
Brief Title: Exercise Strategies to Motivate and Relieve Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU4513
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Chronic Lung Disease; Cardiopulmonary Disease
Keywords: Exercise; Stress; Lung Disease; Music; Podcast
MeSH Terms: conditions — Pulmonary Heart Disease; Motor Activity; Lung Diseases

STUDY DESIGN:
Intervention Model Description: Participants will listen to either self-selected music and then a podcast or podcast and then self-selected music on two consecutive sessions, based on a randomized order.
Who Masked: Participant
Masking Description: Participant is masked to which condition is the experimental intervention of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Condition (Experimental): 3 self-selected music choices to be played during the study
  Interventions: Behavioral: Music Condition
- Podcast Condition (Placebo Comparator): One self-selected podcast choice to be played during the study
  Interventions: Behavioral: Podcast Condition

INTERVENTIONS:
Behavioral: Music Condition — During one of the sessions, participants will listen to music while walking on the treadmill for 10 minutes.
  Arms: Music Condition
Behavioral: Podcast Condition — During one of the sessions, participant will listen to a podcast for 10 minutes while walking on the treadmill.
  Arms: Podcast Condition

SUMMARY:
The goal of this clinical trial is to evaluate exercise strategies that motivate and relive stress in adults with cardiopulomnary conditions. The goals of this study are as follows:

* To explore the feasibility (how easily it can be done) of using self-selected music during exercise training for adults with cardiopulmonary conditions.
* To assess patient satisfaction of self-selected music with exercise for adults with cardiopulmonary conditions.
* To explore the immediate effects of self-selected music on mood and symptoms (shortness of breath and fatigue) compared with listening to a podcast during their exercise training session

Participants will:

* Select 5-7 songs and 1 podcast to listen to during their treatment session
* Walk on the treadmill while either listening to a podcast or music
* Fill out surveys about their mood, symptoms (shortness of breath and fatigue), music/podcast, and exercise

DETAILED DESCRIPTION:
Music2Move aims to assess if tailored music (music choices that are set to a certain beats per minute and are self-selected by the participant) improves mood while exercising in adults with chronic lung diseases, to ultimately motivate them to engage in physical activity more frequently. This trial will be conducted during their pulmonary rehabilitation session for two consecutive sessions. Researchers will flip a coin for a random order of music condition or no music condition for each participant. Researchers will meet with participants before the trial to collect music selections to be played during the pulmonary rehabilitation session. Mood will be assessed every 2 minutes during the trial using the Feeling Scale to examine the effect of tailored music selections on the participants tolerance for exercise and maximal limit exercise exertion during the session. Heart rate, oxygen level, fatigue, and affect (immediate emotional response), measure of breathlessness (feelings of shortness of breath) will also be assessed before and after the trial to examine the affect that tailored music has on physical measures of exercise. The results of this study could aid in finding motivational tools to improve exercise participation and adherence in adults with chronic respiratory disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a cardiopulmonary disease
* Speaks and understands English

Exclusion Criteria:

* Require a hearing aid or have a hearing impairment that interferes with their ability to hear music or use headphones during the study.
* Unable to engage in physical activity due to health conditions including neurological or musculoskeletal diseases.
* Require ≥6 liters of supplemental oxygen during pulmonary rehabilitation sessions.
* Younger than 21 years old.
* Older than 85 years old.
* Have uncontrolled anginal symptoms.
* Unable to exercise on a treadmill.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
FACIT TS-G Score | Day 1 (after the 10 minute walking session)
  The Functional Assessment of Chronic Illness Therapy Treatment Satisfaction General (FACIT TS-G) satisfaction item will be administered to measure participants' satisfaction with the exercise session. This is a 1-item measure with scores range from 0 (poor) to 4 (excellent) with a higher score indicating a better outcome, with a goal of a at least a mean rating of "2."
Total Number of Participants Recruited | Up to 12 weeks
  A priori success benchmark of recruitment efficiency will be the ability to recruit 12 participants for the study.
Percentage of Ecological Momentary Assessment Data Collected | Up to 12 weeks
  A priori success benchmark for collecting ecological momentary assessment data would be to collect ≥80% of mood (Feeling Scale and HR) data as proposed using 2-minute intervals over two, 10-minute exercise sessions.

SECONDARY OUTCOMES:
Score on Positive Items from the Positive and Negative Affect Scale-SF (PANAS-SF) | 10 minutes (after start of walking session)
  The Positive and Negative Affect Scale-SF (PANAS-SF) is a scale that consists of different words that describe feelings and emotions. 10 positive items will be used to assess affect. Scores range from 1-5 with a higher score indicating a a more positive affect. The final score is the sum of the scores for the positive items which ranges from 10 (minimum) to 50 (maximum) with a higher score indicating a more positive affect.
Score on Positive Items from the Physical Activity Affect Scale (PAAS) | 10 minutes (after start of walking session)
  The PAAS is a self-report measure administered during exercise for measuring affect, only the 3 positive items will be administered. Scores range from 0-4 with a "4" indicating a better outcome. The mean of the three positive items on the scale will be taken to calculate the final score which ranges from 0 (minimum) to 4 (maximum), with a higher score indicating a better outcome.
Borg Dyspnea and Fatigue Scale Score | 10 minutes (after start of walking session)
  The Borg Dyspnea and Fatigue Scale are 1-item scales used to measure shortness of breath and fatigue. The score range from 0 (nothing at all) to 10 (very, very severe) with a lower score indicating feeling less of this symptom.
Feeling Scale Score | Up to 10 minutes (after start of walking session)
  The Feeling Scale is 1-item that measures mood ranging from -5 indicating "very bad" to +5 indicating "very good" when asked how they are feeling.
Heart Rate | Up to 10 minutes (after start of walking session)
  Pulsoximeter will be used to measure heart rate.
Dyspnea Anxiety Scale | 10 minutes (after start of walking session)
  Dyspnea Anxiety Scale is a 1-item, 0-100 Visual Analog Scale with scores ranging from 0-100. 0 meaning "not at all anxious" and 100 meaning "extremely anxious."

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Norweg, PhD, Principal Investigator — Columbia University
Locations (1):
- NewYork-Presbyterian Hospital-Columbia Pulmonary Rehabilitation, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No